CLINICAL TRIAL: NCT04351581
Title: Effects of Discontinuing Renin-angiotensin System Inhibitors in Patients With and Without COVID-19
Acronym: RASCOVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-20026484; 2020-001544-26 (EudraCT Number)
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Covid-19
Keywords: COVID-19; RAS; Renin-angiotensin system; Angiotensin II receptor blocker; Angiotensin converting enzyme inhibitor; ARB; ACEi
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: COVID+ Continuation (Experimental): The enrolled patients will continue their prescribed ACEi/ARB in the same dose. The clinicians will be encouraged to continue the medication throughout the hospital admission but it will be permissable for the clinician to stop treatment if necessary e.g. due to hypotension.
  Interventions: Other: Continuation of ACEi/ARB
- B: Covid+ Discontinuation (Experimental): The enrolled patients will discontinue their prescribed ACEi/ARB. If hypertensive treatment is necessary during hospital admission the clinicians will first be encouraged to start non-ACEi/non-ARB treatment; however, if needed it will be possible to start ACEi/ARB again during hospital admission. After study completion (30 days from randomization) the patients will be reminded to seek their generel practitioner to reinitiate ACEi/ARB treatment.
  Interventions: Other: Discontinuation of ACEi/ARB
- C: COVID% Continuation (Experimental): The enrolled patients will continue their prescribed ACEi/ARB in the same dose.
  Interventions: Other: Continuation of ACEi/ARB
- D: COVID% DIscontinuation (Experimental): The enrolled patients will discontinue their prescribed ACEi/ARB. If hypertensive treatment is necessary during the study period clinicians will first be encouraged to start non-ACEi/non-ARB treatment; however, if needed it will be possible to start ACEi/ARB again during the study period. After study completion (30 days from randomization) the patients will be reminded to seek their generel practitioner to reinitiate ACEi/ARB treatment.
  Interventions: Other: Discontinuation of ACEi/ARB

INTERVENTIONS:
Other: Discontinuation of ACEi/ARB — Discontinuation of ACEi/ARB
  Arms: B: Covid+ Discontinuation; D: COVID% DIscontinuation
Other: Continuation of ACEi/ARB — Continuation of ACEi/ARB
  Arms: A: COVID+ Continuation; C: COVID% Continuation

SUMMARY:
Recent data from some of the earliest and worst affected countries of COVID-19 suggest a major overrepresentation of hypertension and diabetes among COVID-19-related deaths and among patients experiencing severe courses of the disease. The vast majority of patients with hypertension and/or diabetes are taking drugs targeting the renin-angiotensin system (RAS) because of their blood pressure-lowering and/or kidney-protective effects. Importantly, the virus causing COVID-19, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) binds to the transmembrane protein angiotensin converting enzyme 2 (ACE2) - an important component of RAS - for host cell entry and subsequent viral replication. ACE2 is normally considered to be an enzyme that limits airway inflammation via effects in RAS and increased ACE2 activity seems to alleviate acute respiratory distress syndrome (ARDS). Importantly, evidence from human studies as well as rodent studies suggests that the inhibition of RAS by angiotensin converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB) leads to upregulation of ACE2, and treatment with ARB leads to attenuation of SARS-CoV-induced ARDS. This is of interest, as the vast majority of deaths from COVID-19 are due to ARDS and expression of ACE2 has previously been shown to be reduced by the binding of SARS-CoV to ACE2. Thus, ACE inhibitors and ARBs have been suggested to alleviate the COVID-19 pulmonary manifestations. In contrast to these notions, concern has been raised that ACE2 upregulation (by RAS-inhibiting drugs) will multiply the cellular access points for viral entry and might increase the risk of severe progression of COVID-19. The multiplied viral entry points could perhaps explain the alarmingly high morbidity and mortality among COVID-19 patients with diabetes and/or hypertension. Thus, a delineation of the role of RAS for the course of COVID-19 is of crucial importance for the management of COVID-19 patients.

Aim:

This randomised clinical trial will investigate whether to continue or discontinue treatment with ACE inhibitors or ARBs in hospitalised patients with COVID-19.

ELIGIBILITY:
Group A and B

Inclusion Criteria:

1. Verified COVID-19
2. Hospital admitted
3. Daily administration of RAS-inhibiting therapy
4. Age 18 years and above
5. Informed consent

Exclusion Criteria:

1. Diagnosed with systolic heart failure (heart failure with reduced ejection fraction)
2. Severe kidney disease; defined by estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m2
3. Severe hypertension; defined by systolic pressure >175 mm Hg and/or diastolic pressure >105 mm Hg
4. Hypotension; defined by systolic pressure <100 mm Hg and/or diastolic pressure <60 mm Hg
5. Non-compliance of RAS-inhibiting therapy; defined as an estimated adherence <80% assessed by a questionnaire in combination with checking the Danish electronic medication system "FMK" (obligatory for clinicians in Denmark to ensure the Danish electronic medication system "FMK" is correct and up-to-date) for redeemed prescriptions in the last six months; in borderline cases, the participant is assumed compatible
6. Pregnancy or breastfeeding
7. Contra indications for receiving ACE inhibitors or ARBs:

   1. Severe liver disease
   2. Hypersensitivity or allergic reactions to the therapy
   3. Angioneurotic edema during previous treatments
   4. Family history of or previous idiopathic angioneurotic edema
   5. Treatment with sacubitril/valsartan or aliskiren

Group C and D:

Inclusion Criteria:

1. Daily administration of RAS-inhibiting therapy
2. Age 18 years and above
3. Informed consent

Exclusion Criteria:

1. Diagnosed with systolic heart failure (heart failure with reduced ejection fraction)
2. Severe kidney disease; defined by estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m2
3. Severe hypertension; defined by systolic pressure >175 mm Hg and/or diastolic pressure >105 mm Hg
4. Hypotension; defined by systolic pressure <100 mm Hg and/or diastolic pressure <60 mm Hg
5. Non-compliance of RAS-inhibiting therapy; defined as an estimated adherence <80% assessed by a questionnaire in combination with checking the Danish electronic medication system "FMK" (obligatory for clinicians in Denmark to ensure the Danish electronic medication system "FMK" is correct and up-to-date) for redeemed prescriptions in the last six months; in borderline cases, the participant is assumed compatible
6. Pregnancy or breastfeeding
7. Contra indications for receiving ACE inhibitors or ARBs:

   1. Severe liver disease
   2. Hypersensitivity or allergic reactions to the therapy
   3. Angioneurotic edema during previous treatments
   4. Family history of or previous idiopathic angioneurotic edema
   5. Treatment with sacubitril/valsartan or aliskiren

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Days alive and out of hospital within 14 days after recruitment (group A vs. group B). | 14 days
  The primary endpoint is days alive and out of hospital within 14 days after recruitment on which a patient satisfies categories 0, 1 or 2 on the eight-category ordinal scale.
  WHO defined Ordinal Scale for Clinical Improvement:
  0. Not hospitalized, no clinical or virological evidence of infection
  1. Not hospitalized, no limitations of activities
  2. Not hospitalized, limitation of activities
  3. Hospitalized, no oxygen therapy
  4. Hospitalized, oxygen by mask or nasal prongs
  5. Hospitalized, non-invasive ventilation or high-flow oxygen
  6. Hospitalized, intubation and mechanical ventilation
  7. Hospitalized, ventilation and additional organ support - pressors, rapid response team (RRT), extracorporeal membrane oxygenation (ECMO)
  8. Death

SECONDARY OUTCOMES:
Key-secondary composite endpoint: Occurrence of worsening of COVID-19 (group A vs. group B) | 30 days
  The key-secondary composite endpoint is the occurrence of worsening of COVID-19 (group A vs. group B) as assessed by when a patient satisfies category 6, 7 or 8 on the ordinal scale within the trial period.
Occurrence and time to occurrence of each of the components of the key-secondary composite endpoint (group A vs. group B) | 30 days
  Occurrence and time to occurrence of each of the components of the key-secondary composite endpoint
Kidney function assessed by plasma creatinine (group A vs. group B) | 30 days
  Kidney function assessed by plasma creatinine
Duration of index hospitalisation (group A vs. group B) | 30 days
  Duration of index hospitalisation
30-day mortality (group A vs. group B) | 30 days
  30-day mortality
Number of days alive during the intervention period (group A vs. group B) | 30 days
  Number of days alive during the intervention period
Number of participants not yet discharged at day 30 (group A vs. group B) | 30 days
  Number of participants not yet discharged at day 30
Number of readmissions after 30 days. (group A vs. group B) | 30 days
  Number of readmissions after 30 days.
Kidney function as assessed by eGFR (group A vs. group B) | 30 days
  Kidney function as assessed by eGFR

OTHER OUTCOMES:
Support for clinical findings via relevant blood markers | 30 days
  To support the clinical findings, blood samples will be analysed for ACE, ACE2, aldosterone, angiotensin II and renin, and expression of ACE, interferon signatures and T cell exhaustion markers.

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital
Locations (2):
- Denmark (2):
  - Department of Medicine, Gentofte Hospital, University of Copenhagen, Hellerup, Capital Region of Denmark
  - Department of Medicine, Herlev Hospital, University of Copenhagen, Herlev, Capital Region of Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang H, Penninger JM, Li Y, Zhong N, Slutsky AS. Angiotensin-converting enzyme 2 (ACE2) as a SARS-CoV-2 receptor: molecular mechanisms and potential therapeutic target. Intensive Care Med. 2020 Apr;46(4):586-590. doi: 10.1007/s00134-020-05985-9. Epub 2020 Mar 3. No abstract available. PMID 32125455
- [Background] Imai Y, Kuba K, Rao S, Huan Y, Guo F, Guan B, Yang P, Sarao R, Wada T, Leong-Poi H, Crackower MA, Fukamizu A, Hui CC, Hein L, Uhlig S, Slutsky AS, Jiang C, Penninger JM. Angiotensin-converting enzyme 2 protects from severe acute lung failure. Nature. 2005 Jul 7;436(7047):112-6. doi: 10.1038/nature03712. PMID 16001071
- [Background] Furuhashi M, Moniwa N, Mita T, Fuseya T, Ishimura S, Ohno K, Shibata S, Tanaka M, Watanabe Y, Akasaka H, Ohnishi H, Yoshida H, Takizawa H, Saitoh S, Ura N, Shimamoto K, Miura T. Urinary angiotensin-converting enzyme 2 in hypertensive patients may be increased by olmesartan, an angiotensin II receptor blocker. Am J Hypertens. 2015 Jan;28(1):15-21. doi: 10.1093/ajh/hpu086. Epub 2014 May 18. PMID 24842388
- [Background] Vuille-dit-Bille RN, Camargo SM, Emmenegger L, Sasse T, Kummer E, Jando J, Hamie QM, Meier CF, Hunziker S, Forras-Kaufmann Z, Kuyumcu S, Fox M, Schwizer W, Fried M, Lindenmeyer M, Gotze O, Verrey F. Human intestine luminal ACE2 and amino acid transporter expression increased by ACE-inhibitors. Amino Acids. 2015 Apr;47(4):693-705. doi: 10.1007/s00726-014-1889-6. Epub 2014 Dec 23. PMID 25534429
- [Derived] Kliim-Hansen V, Gasbjerg LS, Ellegaard AM, Lorentsson HJN, Lynggaard MB, Hagemann CA, Legart C, Mathiesen DS, Sivapalan P, Jensen JS, Vilsboll T, Christensen MB, Knop FK. Protocol for a 30-day randomised, parallel-group, non-inferiority, controlled trial investigating the effects of discontinuing renin-angiotensin system inhibitors in patients with and without COVID-19: the RASCOVID-19 trial. BMJ Open. 2022 Nov 30;12(11):e062895. doi: 10.1136/bmjopen-2022-062895. PMID 36450422